CLINICAL TRIAL: NCT04952870
Title: Exploratory Multicenter Observational Study to Assess the Outcome of Infants With Perinatal SARS-COV-2 Infection and Its Link With the NO Pathway: the Minipuberty Hypothesis
Brief Title: Perinatal Covid-19 Infection, NO Pathway, and Minipuberty
Acronym: miniNO-COVID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_38; 2020-A02122-37 (Other: ID-RCB number, ANSM); grant agreement No 847941 (Other Grant/Funding Number: European Union's Horizon 2020)
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Newborn, Infant, Disease; Neurodevelopmental Disorders
Keywords: Perinatal COVID; newborn; minipuberty; HPG axis; nitric oxide; neurodevelopmental outcome
MeSH Terms: conditions — Disease; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for Genetic analysis Urine for nitrite/nitrates and hormones; Living buccal cells for mRNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 group: Perinatal COVID-19 infection group, including newborns born from COVID-19 infected mothers and newborns with postnatal COVID-19 infections;
- NO group: Newborns admitted in NICU and receiving inhaled NO for respiratory failure
  Interventions: Other: Inhaled NO
- Control group: Newborns admitted in NICU for respiratory failure not receiving iNO and not infected with COVID-19;
  Interventions: Other: routine care

INTERVENTIONS:
Other: Inhaled NO — Newborn or young infants (< 3 months) receiving inhaled NO as part of their treatment for severe respiratory failure
  Groups: NO group
Other: routine care — Patients treated for respiratory failure
  Groups: Control group

SUMMARY:
Some evidence exists that SARS-COV-2 may infect pituitary axis, and therefore may alter hypothalamic function. Whether perinatal COVID-19 is associated with alterations in the maturation of the Hypothalamic-Pituitary-Gonadal (HPG) axis, and specifically with its transient activation occurring during infancy, namely minipuberty, is a major concern. Among the various pathogenic features related to COVID-19, altered minipuberty could be a key factor underlying many multimorbidities later in life, suggesting that they could involve a common causative mechanism that occurs within this short and critical period of time following birth. Altered minipuberty together with NO deficiency seem to be key factors underlying many of these multimorbidities, suggesting that they involve a common causative mechanism that occurs within this short and critical period of time following birth

ELIGIBILITY:
Inclusion Criteria:

* Group 1 : Newborn infants (24 to 41 weeks gestational age) or young infants (< 3 months) admitted at the maternity ward or at the Department of Neonatology at Jeanne de Flandre Hospital, CHU of Lille with perinatal COVID-19 infection defined by:

  * Antenatal COVID-19 infection: pregnant women with positive PCR test at any time of the pregnancy;
  * Post-natal COVID-19 infection: newborn or young infants (< 3 months) with positive PCR test in pharynx or stools as part of their treatment.
* Group 2 : Newborn infants (24 to 41 weeks gestational age) or young infants (< 3 months) admitted at the maternity ward or at the Department of Neonatology at Jeanne de Flandre Hospital, CHU of Lille for severe cardiorespiratory diseases requiring inhaled NO treatment.
* Group 3 : The control group without perinatal COVID-19 infection and no inhaled NO treatment will be matched to the two other groups on age at birth (± 2 weeks of gestation), on postnatal age (± 3 weeks), on respiratory failure (yes/no).
* No inclusion in another ante- or post-natal trial;
* Written consents from both parents.
* Social security affiliation

Exclusion Criteria:

* Preterm birth less than 24 weeks gestational age.
* Severe brain lesions: bilateral and extensive periventricular leukomalacia, intracranial hemorrhage grade 3 or 4;
* One or both of the parents is unable to read or understand French language, or refuse to participate

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborn infants at risk for neurodevelopmental disorders
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The follicle stimulating hormone (FSH) plasma concentrations measured at the postnatal age of 3 months | at the postnatal age of 3 months

SECONDARY OUTCOMES:
The change in reproductive hormones | From the day at inclusion (D0), to Day 2 (48 hours after inclusion), Month 1 and the postnatal age of 3 months
The change in metabolic hormones | From the day at inclusion (D0), to Day 2 (48 hours after inclusion), Month 1 and the postnatal age of 3 months
Rate of negative hearing and olfactive tests | At the postnatal age of 3 months;
Ages and Stages Questionnaire (ASQ-3 ) score | At the corrected age of 9 and 18 months
  The ASQ-3 is a questionnaire aimed to pinpoint developmental progress in children between 1 month to 5.5 years in age. It is parent-centric and is administered through paper and pencil. It takes 10 to 15 minutes to complete. Change in score will be calculated by comparing ASQ-3 scores of FNI and non-FNI participants by measuring across five developmental areas: communication, gross motor, fine motor, problem solving, and personal-social.
Ages and Stages Questionnaire (ASQ-2E) score | At the corrected age of 9 and 18 months
Bayley-III score | at the corrected age of 9 months of age
  The Bayley Scale of Infant and Toddler Development, Third Edition (Bayley III) measures physical, motor, sensory, and cognitive development in babies and young children. The scale encompasses five developmental domains - cognitive, language, motor, social-emotional and adaptive behaviour. The structure of the Bayley-III Scales allows clinicians to administer each of the five scales (cognitive, language-receptive and expressive, motor-fine and gross, social-emotional, and adaptive behaviour) independent of others. Higher scores in each scale indicates more advanced development. Performance is summarised via scaled scores for each subtest, and composite scores for each scale, together with percentile ranks, developmental age equivalents, and growth scores. Discrepancy information is used to determine whether there are significant differences between a child's abilities in the domains measured, and how prevalent these differences are in the norming sample. A total score is not provided.
The time of mutual gaze interactions (versus non-interactive periods) measured by eye-tracking glasses (mother and children) | At the corrected age of 9 months
The specific changes in Nos1-associated genes | From the day at inclusion (D0), Day 2, 1 month and 3 months of age and in buccal cells collected at the postnatal age of 3 months of age.
The specific changes in miRNAs in blood sampled | From the day at inclusion (D0), Day 2, 1 month and 3 months of age and in buccal cells collected at the postnatal age of 3 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent STORME, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- Hop Jeanne de Flandre Chu Lille, Lille, France
- Uri-National and Kapodistrian University of Athens, Athens, Greece